CLINICAL TRIAL: NCT06750120
Title: An Integrated Intervention to Address the Double Burden of Malnutrition in Guatemala
Brief Title: Addressing the Double Burden of Malnutrition in Guatemala
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Wuqu' Kawoq, Maya Health Alliance (Other); Instituto de Nutricion de Centroamerica y Panama (INCAP) (Unknown); University of Michigan (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Peter J. Rohloff, M.D.,Ph.D., Associate Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P003339
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Maternal Obesity Complicating Pregnancy, Birth,or Puerperium; Child Malnutrition
Keywords: Guatemala; stunting; maternal obesity; food supplementation; lifestyle counseling
MeSH Terms: conditions — Child Nutrition Disorders; Growth Disorders; Pregnancy in Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Arm (Experimental): Two intervention components will be provided from enrollment through 12 months postpartum:
  1. Monthly household food rations providing 5 daily food groups and a mean of 165 kcal/per capita/day
  2. Behavioral counselling by frontline health workers to promote healthy gestational weight gain and post partum weight loss.
  Participants will also receive enhanced usual care as described for the active comparator arm.
  Interventions: Dietary Supplement: Family food ration; Behavioral: Optimal weight counseling; Other: Enhanced Usual Care
- Enhanced Usual Care Arm (Active Comparator): The comparator will be enhanced usual care alone, which will include:
  Usual care: free standard pregnancy, postnatal, and infant care through Ministry of Health services.
  Enhancements to usual care: Participants in both arms will be enrolled in Maya Health Alliance's free care navigation program. In this program, navigators accompany patients to clinical visits at national hospitals, provide interpretation, and cover emergency transportation cost.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Dietary Supplement: Family food ration — Monthly household food rations providing 5 daily food groups and a mean of 165 kcal/per capita/day
  Arms: Intervention Arm
Behavioral: Optimal weight counseling — Counseling on health gestational weight gain and post partum weight loss
  Arms: Intervention Arm
Other: Enhanced Usual Care — Enhanced usual care includes
  1. Usual care: free standard pregnancy, postnatal, and infant care through Ministry of Health services.
  2. Enhancements to usual care: Participants in both arms will be enrolled in Maya Health Alliance's free care navigation program. In this program, navigators accompany patients to clinical visits at national hospitals, provide interpretation, and cover emergency transportation cost.

SUMMARY:
Globally, populations are experiencing increases in the double burden of malnutrition, commonly defined as maternal overweight/obesity and child stunting in the same household. In this study, we will evaluate how a combined intervention including both counseling for healthy weight in mothers and food supplementation for families can reduce the double burden of malnutrition in rural Guatemala.

DETAILED DESCRIPTION:
Globally, populations are experiencing increases in diseases attributable to overnutrition, but child undernutrition also persists at high levels. This "double burden of malnutrition" commonly appears as maternal overweight/obesity and child stunting in the same household. Poor nutrition during the critical life stages of the pregnancy, the postpartum period, and early childhood increases life-long risk for nutrition-related non-communicable diseases such as diabetes, hypertension, and dyslipidemia for both mother and child. Evidence-based interventions exist that promote optimal weight gain during pregnancy and postpartum weight loss or prevent undernutrition among children, but little is known about implementing them as integrated, scalable, intergenerational, affordable, and equity-focused solutions. The overall goal of this project is to assess the effectiveness, implementation, and cost-effectiveness of an integrated intervention to reduce the double burden of malnutrition among pregnant/postpartum women and their children. We will conduct a type 1 hybrid effectiveness-implementation trial in rural Guatemalan Indigenous communities that have among the world's highest prevalence of the double burden of malnutrition. Our project will have three parts. In Part 1, we will conduct an individually randomized hybrid type 1 effectiveness-implementation trial with 766 pregnant mothers and their children, including both food supplementation and counselling to optimize mothers' gestational weight gain and limit postpartum weight retention. Our primary evaluation will focus on maternal weight and child length at 12 months after birth. In Part 2, we will assess barriers and facilitators to implementation of the integrated DBM intervention and develop strategies to promote widespread implementation. In Part 3, we will conduct an economic evaluation on the integrated nutrition intervention. To our knowledge, this aim will generate the first evidence of costs and cost-effectiveness of interventions to address DBM at the household level, providing crucial information to policymakers and stakeholders for future implementation and budgeting. Overall, this project will generate globally relevant implementation evidence on interventions for the double burden of malnutrition. Results will have implications for nutrition and NCD policy not only in Guatemala but also globally. A major feature of the project is a focus on pragmatism and equity, working to enroll the most vulnerable families from rural Guatemala who stand most to benefit from the intervention but who are commonly excluded from clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women < 28 weeks gestation,
* aged >=16years
* subject willing and able to provide informed consent

Exclusion Criteria:

* Prior self-reported history of pre-eclampsia, gestational or pregestational diabetes
* >= 28 weeks gestation at enrollment visit
* Gestational or pregestational diabetes will be defined by self-report or hemoglobin A1c (HbA1c) ≥6.5% at enrollment.

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1532 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Maternal weight | 12 months post partum
  Difference in mean maternal weight (kg) between arms at 12 mo. postpartum
Infant length for age Z score | 12 months post partum
  Between group difference in mean child lengthforage z score at 12 mo. using WHO growth standards.

SECONDARY OUTCOMES:
Adequacy of maternal gestational weight gain | 1 Month preceding delivery
  Difference in initial and final pregnancy weight using IOM cut points, means compared between arms. Prepregnancy BMI will be estimated using self-reported prepregnancy weight and enrollment height.
Postpartum maternal waist to hip ratio | 6 and 12 month postpartum
  Difference in waist to hip ratio between arms at 6 and 12 mo. postpartum
Maternal physical activity | 12 months postpartum
  Global Physical Activity Questionnaire. Means compared between arms.
Maternal dietary diversity | 36 weeks gestation and 12 months postpartum
  Minimum Dietary Diversity for Women tool,which is a validated proxy measure of micronutrient adequacy among cohorts of reproductive-age women. Proportions compared between arms
Household food insecurity | 36 weeks gestation and 12 months postpartum
  Food Insecurity Experience Scale. Means compared between arms
Maternal Hemoglobin | 12 months postpartum
  WHO anemia cut points will be adjusted for elevation. Proportion of anemia compared between arms.
Maternal health-related quality of life | 36 weeks gestation and 12 months postpartum
  WHOQOL-BREF tool; means compared between arms.
Neonatal and infant mortality | 12 months postpartum
  Adjudicated by study staff using facility records and/or verbal autopsy. Final rates compared between arms at study exit (12 mo post partum).
Infant hemoglobin | 12 months of age
  WHO anemia cut points will be adjusted for elevation. Proportion of anemia compared between arms.
Global child development | 12 months of age
  Caregiver Reported Early Child Development Instruments (CREDI) long form, which has been validated in Indigenous populations in Guatemala. Mean age-adjusted Z scores compared between arms

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rohloff, MD PhD, Principal Investigator — Brigham and Women's Hospital; Manuel Ramirez, MD PhD, Principal Investigator — Institute of Nutrition of Central America and Panama

IPD SHARING:
Plan to Share IPD: Yes
De-identified databases containing all study data, including survey and clinical findings and coded variables
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning at the time of publication of the main study paper or completion of primary study data collection and cleaning, whichever comes first, with no end date
Access Criteria: All data will be stored and accessible through the NICHD DASH repository, following standard procedure for that repositoiry, requiring the completion of a Data Use Agreement which prohibits any redistribution or attempts to re-identify research participants.

REFERENCES:
- [Background] Popkin BM, Corvalan C, Grummer-Strawn LM. Dynamics of the double burden of malnutrition and the changing nutrition reality. Lancet. 2020 Jan 4;395(10217):65-74. doi: 10.1016/S0140-6736(19)32497-3. Epub 2019 Dec 15. PMID 31852602